CLINICAL TRIAL: NCT06342674
Title: Effect of Breast Milk Circadian Properties on Infant Growth Parameters and Nutrient Absorption in Preterm Newborns
Brief Title: Effect of Breast Milk Circadian Properties on Infant's Growth Parameters and Absorption of Nutrients
Acronym: The
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, dilek menekşe, Assistant professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Nejla CANBULAT ŞAHİNER
Record Dates: First submitted 2024-01-20; First posted 2024-04-02 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Breast Feeding; Breast Milk Collection
Keywords: Breast milk; circadian rhythm; growth; preterm; newborn
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression; Premature Birth

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Single (participant) blinding was used in the study. For this purpose, it was not stated which group the participating mothers were in the research, but they were informed about the procedure to be performed. Therefore, a separate informed consent form was prepared for each group. Statistician blinding will also be applied. While coding the research data, the research group will be coded as A and B, and the statistician will be prevented from knowing which letter represents which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): While the mothers' babies are in the neonatal intensive care unit, the babies in the circadian rhythm group will be fed by taking into account the date and day/night practice. The milk that the mother expresses at night will be given to her baby at night, and the milk that she expresses during the day will be used for daytime feeding. Milk expressed 24 hours a day is delivered to the baby in 4 time periods (06:00-12:00, 12:00-18:00, 18:00-24:00, 24:00-06:00) in coordination with the time it is expressed. It is planned to be given (Italianer et al., 2020).For example, the milk expressed at 02:00 at night on 15.08.2023 and at 05:00 at night on 16.08.2023 will be given to the baby first with the milk of the previous date of 15.08.2023, in the period of 24:00-06:00 at night. Breast milk will be given according to both date and day/night milk concept.
  Interventions: Other: Giving breast milk to the newborn according to the circadian rhythm
- Control Groups (Experimental): In the control group, the condition of "expressed milk is given first", which is used in routine practice, will be fulfilled, regardless of the day and night characteristics of expressed breast milk. The routine practice of the clinic will continue.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Giving breast milk to the newborn according to the circadian rhythm — It is the delivery of milk expressed by the newborn's mother during the neonatal intensive care unit, in accordance with the time of expression. Breast milk follows the circadian rhythm, that is, the milk the mother expresses at night will be given to her infant at night, and the milk she expresses during the day will be given to her infant during the day
  Arms: Experimental Group
Other: Usual care — Newborns in the control group will be given expressed milk first, in line with the routine practice of the clinic
  Arms: Control Groups

SUMMARY:
The most ideal method for providing breast milk is breastfeeding. However, it may be necessary to express breast milk for reasons such as the newborn being in an intensive care unit, the mother being hospitalized for any reason, or the mother starting to work. The content of breast milk varies according to gestational age and stages of lactation. However, it varies from day to day depending on the infant's needs. In recent literature, it is emphasized that the content of breast milk (carbohydrates, fats, proteins, vitamins, trace elements, etc.) varies according to circadian variation. In the literature review, no national or international study was found indicating whether the circadian properties of breast milk have an effect on the infant's growth parameters. This study was designed as a randomized controlled experimental study to determine the effect of the circadian properties of breast milk on the growth parameters of the infant and the absorption levels of nutrients by the baby in preterm newborns.

no effect on the infant's growth parameters and nutrient absorption levels by the infant.

Hypothesis 1 (H1): Feeding preterm newborns with breast milk according to the circadian rhythm has an effect on the weight of the infants.

Hypothesis 2 (H2): Feeding preterm newborns with breast milk according to the circadian rhythm has an effect on the height of the infants.

Hypothesis 3 (H3): Feeding preterm newborns with breast milk according to the circadian rhythm has an effect on the head circumference of the infants.

Hypothesis 4 (H4): Feeding preterm newborns with breast milk according to the circadian rhythm has an effect on the absorption levels of vitamins and trace elements measured in the infants' breast milk.

DETAILED DESCRIPTION:
Breast milk is an ideal and unique food with excellent content for the healthy growth and development of both term and preterm babies. Breast milk, which is considered the "Gold Standard" in term and preterm baby nutrition, has a complex, lively and dynamic structure. The content of breast milk varies from day to day and according to the gestational age, stages of lactation, and the baby's needs. These differences indicate that breast milk is a unique food.

Breast milk contains many complex nutrients, and while the amount of some nutrients varies depending on the mother's diet, lactation day and duration, some nutrients remain at relatively constant levels. Breast milk contains macronutrients (carbohydrates, proteins, fats), micronutrients (vitamins, trace elements and electrolytes) and bioactive factors (various hormones, immune factors and other bioactive factors). In recent years, the difference in the content of breast milk according to circadian variation has been evaluated. In studies examining breast milk content according to circadian variation, it was stated that total carbohydrate concentration did not show circadian change.It has been determined that the fat concentrations in breast milk, which are necessary for the growth and development of the baby, indicate the existence of circadian variation. However, there are different results in element and vitamin studies. In cases where breast milk should be given by expressing, not giving milk in accordance with the circadian rhythm may disrupt the developing circadian rhythms of babies, potentially causing sleep problems and decreased physiological harmony with their parents/environment. This situation may negatively affect the baby's growth and development and endanger its health. In light of this information; The study was planned to determine the effect of the circadian properties of breast milk on the growth parameters of the baby and the absorption levels of nutrients by the baby in preterm newborns.

ELIGIBILITY:
Inclusion Criteria:

* The mother is healthy (without a history of preeclampsia, hypertension, diabetes, hepatitis B or C, HIV, tuberculosis, mastitis or oncological disease)
* The mother's birth is 32-34 between weeks of gestation
* The mother does not follow a special diet
* The mother is not a vegetarian
* The mother does not smoke
* The mother must have a body mass index within normal limits (BMI = 18.50-24.99) (WHO, 2022b)
* Income must be at or above the monthly minimum wage
* The mother cannot breastfeed her baby and routinely expresses her own milk every three hours.
* The mother expresses her milk with a milking machine (milking will be done with the same brand device and the same level of suction power).
* The baby is in the neonatal intensive care unit
* Feeding the infant by gavage and oral method

  *In order for the preterm newborn to be fed effectively and safely orally, it is necessary for the preterm baby to be able to coordinate sucking-swallowing as well as breathing (Tian et al., 2015). Gavage feeding is a priority in babies who have this coordination (TND, 2018). In babies who have the coordination of sucking, swallowing and breathing, oral feeding will be started after an assessment of readiness for oral feeding will be made.
* Full enterally fed babies
* The infant does not have a health problem that requires surgical treatment
* 10th-90th percentile curves according to the infant's gestational age. percentile (those with normal birth weight for gestational age: Appropriate for Gestational Age -AGA)

Exclusion Criteria:

* The mother receives medication (antibiotics, etc.) treatment
* Interruption of the mother's milk during the working period
* Low birth weight of the baby according to the intrauterine growth curve
* Feeding the baby with formula
* Total parenterally fed babies
* The baby has a small birth weight for the gestational age (Small for Gestational Age - SGA) and a baby with a large birth weight for the gestational age (LGA).

Criteria for Exclusion from the Study;

* The mother received medication (antibiotics, etc.) during the data collection process.
* The mother does not want to continue
* Respiratory problems, hypoglycemia, hyperbilirubinemia, etc. in preterm babies. occurrence of various problems

Ages: 32 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the newborn's body weight in the study and control groups Evaluation of the newborn's body weight in the study and control groups Evaluation of the newborn's body weight in the study and control groups | Difference between the first measurement before application (in birth) and the body weight measurement at discharge (an average of one month after birth)
  A calibrated scale, capable of weighing accurately to 10 grams, will be used to measure the weight of infants. During the process, a disposable cover will be placed on the scale to be measured, and the scale will be set to "0". The baby's clothes will be removed and the baby will be measured naked except for the dry diaper. If a dry diaper is left, the weight of the diaper will be deducted from the child's body weight. Measurements will be made once every two days for four weeks.
Evaluation of the baby's height measurements in the study and control groups | Difference between the first measurement before application (in birth)and the body height measurement at discharge (an average of one month after birth)
  A height meter will be used to measure the height of babies. Height measurements of babies will be made in the supine position. If the baby has any booties, shoes or hat, they will be removed and the measurement will be performed. Care must be taken to ensure that the ground on which the measurement will be made is hard and horizontal. The baby's head will be kept in contact with the fixed board, and the other will be measured by sliding the moving part to the baby's sole. Measurements will be made once every two days for four weeks.
Evaluation of the baby's head circumference in the study and control groups | Difference between the first measurement before application (in birth) and head circumference measurement at discharge (an average of one month after birth)
  A tape measure will be used to measure babies' head circumference. Measurement of the baby's head circumference; It will be measured by passing the non-flexible tape measure over the most protruding occiput bone at the back of the head, over the ears on the side, and over the eyebrows in front. Measurements will be made once every two days for four weeks

SECONDARY OUTCOMES:
Evaluation of nutritional absorption of infants in the study and control groups | Difference between first measurement (postpartum) (in birth) and second measurement (at discharge) (an average of one month after birth)
  25-30 ml of breast milk will be used for all milk analyses. Breast milk melatonin hormone levels will be analyzed by Enzyme Plate Reader by taking 50 µl of milk and using the ELISA kit.Serum content parameters of the mother and the newborn will be evaluated. During the routine practice of the clinic, blood samples from the mother and the baby will be taken after birth (for the first time) and at discharge (approximately 1 month later). After the blood samples are used for laboratory analysis in accordance with the requests of the clinic, the remaining samples will be taken from the laboratory (1 ml), sampled separately for serum, vitamin and trace element analyzes and transferred to storage bottles with a pipette. Nutrient analyzes will be performed by Inductively Coupled Plasma-Optical Emission Spectrometry and High Performance Liquid Chromatography

CONTACTS AND LOCATIONS:
Overall Officials: Nejla Canbulat Şahiner, Prof.Dr., Study Director — Karamanoğlu Mehmet Bey University; Ayşe Sonay Türkmen, Prof. Dr., Principal Investigator — Karamanoğlu Mehmet Bey University; Dilek Menekşe, Asst. prof., Principal Investigator — Sakarya University; Hacer Sibel Karapınar, Assoc. Prof., Principal Investigator — Karamanoğlu Mehmet Bey University; Murat Konak, Assoc. Prof., Principal Investigator — Selcuk University; Havvanur Bayam, Nutritionist, Principal Investigator — Selcuk University
Locations (1):
- Karamanoğlu Mehmet Bey University, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Menekşe, D., Çınar, N.2017. "Çoğul Bebeklerde Emzirme", Turkiye Klinikleri J Pediatr Nurs-Special Topics. 3,2, 91-103.
- [Background] Italianer MF, Naninck EFG, Roelants JA, van der Horst GTJ, Reiss IKM, Goudoever JBV, Joosten KFM, Chaves I, Vermeulen MJ. Circadian Variation in Human Milk Composition, a Systematic Review. Nutrients. 2020 Aug 4;12(8):2328. doi: 10.3390/nu12082328. PMID 32759654
- [Background] Gidrewicz DA, Fenton TR. A systematic review and meta-analysis of the nutrient content of preterm and term breast milk. BMC Pediatr. 2014 Aug 30;14:216. doi: 10.1186/1471-2431-14-216. PMID 25174435
- [Background] Sahin S, Ozdemir T, Katipoglu N, Akcan AB, Kaynak Turkmen M. Comparison of Changes in Breast Milk Macronutrient Content During the First Month in Preterm and Term Infants. Breastfeed Med. 2020 Jan;15(1):56-62. doi: 10.1089/bfm.2019.0141. Epub 2019 Nov 25. PMID 31765240
- [Background] Ovalı, F. 2018. "0-1 yaş bebeklerde vitamin, mineral ve eser element desteği", Klinik Tıp Pediatri Dergisi, 10,1, 1-6.
- [Background] McNaughton L, Davies P. The effects of a 16 week aerobic conditioning program on serum lipids, lipoproteins and coronary risk factors. J Sports Med Phys Fitness. 1987 Sep;27(3):296-302. No abstract available. PMID 3431112
- [Background] Moran-Lev H, Mimouni FB, Ovental A, Mangel L, Mandel D, Lubetzky R. Circadian Macronutrients Variations over the First 7 Weeks of Human Milk Feeding of Preterm Infants. Breastfeed Med. 2015 Sep;10(7):366-70. doi: 10.1089/bfm.2015.0053. Epub 2015 Jul 29. PMID 26222826
- [Background] Hollanders JJ, Kouwenhoven SMP, van der Voorn B, van Goudoever JB, Rotteveel J, Finken MJJ. The Association between Breastmilk Glucocorticoid Concentrations and Macronutrient Contents Throughout the Day. Nutrients. 2019 Jan 24;11(2):259. doi: 10.3390/nu11020259. PMID 30682836
- [Background] Hampel D, Shahab-Ferdows S, Islam MM, Peerson JM, Allen LH. Vitamin Concentrations in Human Milk Vary with Time within Feed, Circadian Rhythm, and Single-Dose Supplementation. J Nutr. 2017 Apr;147(4):603-611. doi: 10.3945/jn.116.242941. Epub 2017 Feb 15. PMID 28202638
- [Background] Hahn-Holbrook J, Saxbe D, Bixby C, Steele C, Glynn L. Human milk as "chrononutrition": implications for child health and development. Pediatr Res. 2019 Jun;85(7):936-942. doi: 10.1038/s41390-019-0368-x. Epub 2019 Mar 11. PMID 30858473